CLINICAL TRIAL: NCT03218735
Title: Early Term Delivery Versus Expectant Management of the Large for Gestational Age Fetus (TEAM LGA Trial)
Brief Title: Early Term Delivery Versus Expectant Management of the Large for Gestational Age Fetus
Acronym: TEAM LGA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: It was discovered that the patient population would not be large enough to adequately recruit.
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Harris Health System, Lyndon B Johnson Hospital obstetrics and gynecology clinic (Unknown)
Responsible Party: Principal Investigator, Bahaeddine M Sibai, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC-MS-17-0110
Record Dates: First submitted 2017-07-12; First posted 2017-07-17 (Actual); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Macrosomia, Fetal; Labor Induction
Keywords: large for gestational age fetal growth
MeSH Terms: conditions — Fetal Macrosomia | interventions — Pregnancy; Parturition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Labor induction at 37.0 weeks to 37.6 weeks of gestation (Experimental): Diagnosis of LGA with induction at 37 weeks 0 days of gestation to 37 weeks and 6 days
  Interventions: Procedure: Labor induction at 37.0 weeks to 37.6 weeks of gestation
- Expectant monitoring and delivery (Active Comparator): Diagnosis of LGA with expectant monitoring and delivery as indicated by standard obstetric practices
  Interventions: Procedure: Expectant monitoring and delivery

INTERVENTIONS:
Procedure: Labor induction at 37.0 weeks to 37.6 weeks of gestation — Diagnosis of LGA with induction at 37 weeks 0 days of gestation to 37 weeks and 6 days
  Arms: Labor induction at 37.0 weeks to 37.6 weeks of gestation
Procedure: Expectant monitoring and delivery — Diagnosis of LGA with expectant monitoring and delivery as indicated by standard obstetric practices
  Arms: Expectant monitoring and delivery

SUMMARY:
The purpose of this study is to compare the incidence of composite neonatal morbidity and birthweight >4500 grams among uncomplicated large for gestational age (LGA) fetal growth at delivered 37 weeks versus expectant management.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Plan for vaginal delivery. Patients with prior cesarean section are eligible if they are planning for a trial of labor after cesarean section.
* Gestational age 34 weeks 0 days to 37 weeks 0 days at time of enrollment
* Dating of pregnancy by last menstrual period consistent with an ultrasound, ultrasound <21 weeks and 6 days of gestation, or known date of conception in the setting of in vitro fertilization
* No known major anomalies (anomalies requiring surgery antenatally or in the neonatal period, anomalies not compatible with life as determined by the physician)
* LGA defined as estimated fetal weight (EFW) > 90th percentile by Hadlock formula but <4500 grams

Exclusion Criteria:

* Pre-gestational diabetes or gestational diabetes on medication (oral or insulin, excluding metformin)
* Planned cesarean delivery
* Polyhydramnios
* Known major fetal anomalies
* Multiple gestation or selective reduction of multiple gestation after 14 weeks
* Previous stillbirth at term
* Indications for delivery at <39 weeks. Common examples include:
* Placenta previa
* Placenta accreta
* Vasa previa
* History of classical cesarean section or myomectomy
* Human immunodeficiency virus (HIV)
* Oligohydramnios (low amniotic fluid, defined as maximum vertical pocket <2.0cm)
* High-risk pregnancy as determined by the physician. Common examples include:
* Pre-gestational diabetes or gestational diabetes on medication
* Chronic hypertension on medication
* Maternal cardiac disease
* Asthma requiring oral steroids during pregnancy
* Chronic renal disease
* Antiphospholipid syndrome
* Hyperthyroidism
* Prior stillbirth
* Systemic lupus erythematous
* Hemoglobinopathies such as sickle cell disease

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07-12 (Actual); Primary Completion 2019-07-01 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
Number of children presenting with CNM | Up to 6 weeks after delivery
  Composite neonatal morbidity (CNM) is any of the following: Apgar score <5 at 5 minutes, seizure, fracture of skull, humerus, or clavicle, neonatal brachial plexus palsy, facial nerve palsy, oxygen supplementation >4 hours, CPAP >2 hours, mechanical ventilation, or death before discharge or IUFD.
Number of children with birthweight above 4500 grams | Immediately at birth

SECONDARY OUTCOMES:
Number of women presenting with CMM | Up to 6 weeks after delivery
  Composite maternal morbidity (CMM) is any of the following: chorioamnionitis, shoulder dystocia, 3rd or 4th degree laceration or episiotomy, transfusion of blood products, endometritis, wound infection or separation, deep venous thrombosis, pulmonary embolism, admission to the intensive care unit, or death. Rates of cesarean section as well as indications in each group will also be evaluated.
Number of children delivered by cesarean section | Immediately at birth
Number of children admitted to NICU | Up to 6 weeks after delivery
  NICU is neo-natal intensive care unit

CONTACTS AND LOCATIONS:
Overall Officials: Baha M Sibai, MD, Principal Investigator — The University of Texas Health Science Center, Houston